CLINICAL TRIAL: NCT06375590
Title: NavIIcusp: Bicuspid Aortic Valve Stenosis With Navitor Platform International Experience
Status: Not yet recruiting | Type: Observational
Sponsor: Didier TCHETCHE (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor-Investigator, Didier TCHETCHE, Head of structural heart disease program, Clinique Pasteur
Organization: Clinique Pasteur (Other)
Other Study IDs: 2024-NavIIcusp
Record Dates: First submitted 2024-04-07; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Bicuspid Aortic Valve
Keywords: Bicuspid aortic valve; TAVI; Navitor
MeSH Terms: conditions — Bicuspid Aortic Valve Disease | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Bicuspid aortic valve: Treated with Navitor platform
  Interventions: Device: Transcatheter Aortic Valve Implantation

INTERVENTIONS:
Device: Transcatheter Aortic Valve Implantation — Transcatheter treatment of bicuspid stenosis with the Navitor platform
  Other Names: Transcatheter Aortic Valve Replacement

SUMMARY:
The aim of this prospective registry is to evaluate the clinical impact of the new Navitor prosthesis (Abbott, Minneapolis, MN, USA) in BAV and evaluate both the main sizing methods (the classical annular or the supra-annular with ICD measurement at 4 mm above the virtual basal ring).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. NYHA ≥ 2 and/or syncope and/or angina.
3. Symptomatic severe calcified aortic stenosis with AVA < 1 cm2 AND peak velocity > 4 m/s or mean gradient > 40 mmHg or DVI < 0.25'.
4. Patient judged by the Heart Team as indicated for TAVI.
5. Anatomical suitability for transfemoral-TAVI with Navitor, based on MSCT assessment.
6. Estimated life-expectancy > 1 year.

Exclusion Criteria:

1. Age < 18 years
2. Asymptomatic patients
3. Estimated life expectancy < 1 year
4. Pure aortic regurgitation.
5. LVEF < 20%
6. No baseline MSCT evaluation.
7. Unsuitable aortic root anatomy for Navitor.
8. Unsuitable peripheral vasculature for transfemoral Navitor.
9. Type 2 bicuspid aortic valve
10. Excessive leaflet calcifications
11. Moderate or severe raphe calcifications
12. Severe LVOT calcifications
13. Perimeter-derived annular dimension exceeding IFU recommendation
14. Dilated ascending aorta >45 mm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients presenting with severe and symptomatic bicuspid aortic valve stenosis or mixed disease
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
30-day device success (Rate) | 30-day
  as indicated in the VARC-3 criteria

SECONDARY OUTCOMES:
1 year at least moderate bioprosthetic valve deterioration | 1-year
  defined as increase in mean transvalvular gradient ≥10 mmHg resulting in mean gradient ≥20 mmHg with concomitant decrease in EOA ≥0.3 cm2 or ≥25% and/or decrease in Doppler velocity index ≥0.1 or ≥20% compared with echocardiographic assessment performed 1-3 months post-procedure, OR new occurrence or increase of ≥1 grade of intra-prosthetic AR resulting in ≥ moderate AR
1 year severe patient-prosthesis mismatch | 1-year
  defined as EOAi < 0.65 cm2/m2
30 days and 1 year all-cause and cardiovascular mortality | 1-year
30 days and 1 year stroke | 1-year

CONTACTS AND LOCATIONS:
Overall Officials: Didier Tchétché, MD, Principal Investigator — Clinique Pasteur
Locations (1):
- Clinique Pasteur, Toulouse, Occitanie, France

IPD SHARING:
Plan to Share IPD: Undecided
Mutual anonymized database. Substudies anticipated.